CLINICAL TRIAL: NCT02367391
Title: Pilot Randomized Trial of an Automated Smoking Cessation Intervention Via Mobile Phone Text Messages as an Adjunct to Varenicline in Primary Care
Brief Title: Penn State TXT2Quit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 41720
Record Dates: First submitted 2015-02-13; First posted 2015-02-20 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Nicotine Dependence, Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Text Messages (Experimental)
  Interventions: Behavioral: Motivational Text Messages
- Control (Sham Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Motivational Text Messages — Usual care plus motivational text messages sent via Mobile Phone. All participants receive the active medication, Varenicline.
  Arms: Motivational Text Messages
Behavioral: Control — Usual Care. All participants receive the active medication, Varenicline.
  Arms: Control

SUMMARY:
This study is evaluating the feasibility and short term smoking cessation outcomes of an automated smoking cessation intervention delivered via mobile phone text messaging as an adjunct to Varenicline in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Smoke >4 cigarettes/day for at least 6 months
* Age 21+
* Want to quit and ready to try in next 30 days
* Willing to quit all forms of tobacco (including e-cigs)
* Willing to use Chantix to try to quit
* Have a cell phone able to receive text messages
* Willing to attend 3 visits and use varenicline for smoking cessation
* Plan to live in local area for next 6 months
* Read and write in English
* Women not pregnant and taking steps to avoid
* Able to understand and willing to sign consent

Exclusion Criteria:

* History of allergic reaction or other adverse event while using varenicline
* Used a smoking cessation aid/medicine in past 1 month (including e-cigs)
* Currently pregnant or nursing
* Does not have a mobile phone that can send and receive text messages or unwilling to receive study texts
* Uncontrolled serious mental illness or substance abuse or inpatient treatment for these in the past 6 months
* Uses non-cigarette tobacco products and does not plan to quit all tobacco.
* Has a history of kidney problems or receives dialysis
* Had any thoughts that they would be better off dead or of deliberate self-harm in the prior 4 weeks
* Had a heart attack in the past 4 weeks
* Mental conditions that would prohibit the participant from completing the protocol

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Yingst JM, Veldheer S, Hrabovsky S, Hammett E, Nicholson J, Berg A, Foulds J. Pilot Randomized Trial of an Automated Smoking Cessation Intervention via Mobile Phone Text Messages as an Adjunct to Varenicline in Primary Care. J Health Commun. 2018;23(4):370-378. doi: 10.1080/10810730.2018.1453890. Epub 2018 Mar 26. PMID 29578832

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Motivational Text Messages | Control
Started | 76 | 76
Completed | 74 | 76
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Text Messages | Control | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.3) | 44.5 (11.6) | 45.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 54 | 99
  Male | 29 | 22 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 65 | 66 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 74 | 76 | 150

OUTCOME MEASURES:

1. Primary Outcome: Point Prevalence of 7-day Tobacco Abstinence Biochemically Validated by Exhaled CO < 10ppm at Visit 3 (12 Weeks After Target Quit Day)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 74 | 76
Participants | 23 | 23

2. Primary Outcome: Sustained Abstinence at the 12-week Follow up
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 74 | 76
Participants | 6 | 9

3. Primary Outcome: Number of Days of Varenicline Use
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 74 | 76
days | 55.4 (37.2) | 55.7 (35.5)

4. Primary Outcome: Number of Active Smoking Cessation Activities Used
Description: Number of activities completed out of 6
Time Frame: 12 weeks
Population: This data is presented for only participants who showed to Visit 2.
Measure: Mean (Standard Deviation); unit: activities
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 60 | 62
activities | 4.5 (1.3) | 4.0 (1.5)

5. Secondary Outcome: Continuous Lapse-free Tobacco Abstinence From 4 Weeks to 12 Weeks, Biochemically Validated at Visit 2 and Visit 3.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 74 | 76
Participants | 6 | 9

6. Secondary Outcome: Time (in Days) to Relapse After the Target Quit Day
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 74 | 76
days | 16.0 (28.9) | 16.5 (30.6)

7. Secondary Outcome: Total Score on the Positive Smoking Cessation Activities Measure
Description: Total score for 6 items (scored 0-3). Total score range 0-18.
Time Frame: 12 weeks
Population: This data is presented for only participants who showed to Visit 2.
Measure: Mean (Standard Deviation); unit: activities
Arm/Group | Motivational Text Messages | Control
Number analyzed (Participants) | 60 | 62
activities | 10.5 (3.8) | 9.1 (4.2)

ADVERSE EVENTS:
Arm/Group | Motivational Text Messages | Control
Serious Adverse Events (participants affected / at risk) | 1/74 | 2/76
Other Adverse Events (participants affected / at risk) | 39/74 | 33/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Text Messages (N=74) | Control (N=76)
Development of Diabetes (Endocrine disorders) | 1 (1) | 0 (0)
Gallbladder Surgery (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Motivational Text Messages (N=74) | Control (N=76)
Nausea (Gastrointestinal disorders) | 11 | 11
Vivid or Unusual Dreams (Psychiatric disorders) | 8 | 9
Nicotine Withdrawal Symptoms (Psychiatric disorders) | 10 | 11
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Thoughts of death (Psychiatric disorders) | 1 | 1
Excessive Sweating (Endocrine disorders) | 1 | 1
Increased mucus production in eye (Eye disorders) | 1 | 0
Migraines (Nervous system disorders) | 1 | 0
Increased Salivation (Gastrointestinal disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Abdominal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Ringing in ears (Ear and labyrinth disorders) | 1 | 0
Vomitting (Gastrointestinal disorders) | 1 | 0
Chest Pain (Cardiac disorders) | 0 | 1
Skin Peeling (Skin and subcutaneous tissue disorders) | 1 | 0
Increase in hot flashes (Reproductive system and breast disorders) | 1 | 0
Coughing up blood (Gastrointestinal disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Stomach Pain (Gastrointestinal disorders) | 0 | 1
Balance Problems (Ear and labyrinth disorders) | 1 | 0
Drug/Alcohol Rehab (Social circumstances) | 1 | 0
Hysterectomy (Reproductive system and breast disorders) | 1 | 0
Pregnancy (Reproductive system and breast disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No